CLINICAL TRIAL: NCT01403662
Title: A Pilot, Open-label, 8-Week Study Evaluating the Efficacy, Safety, and Tolerability of Adjunctive Minocycline for the Treatment of Bipolar Depression
Brief Title: Evaluating the Efficacy of Adjunctive Minocycline for the Treatment of Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Roger McIntyre, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3420337
Record Dates: First submitted 2011-07-18; First posted 2011-07-27 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Bipolar Disorder; Bipolar Depression; Bipolar I Depression; Bipolar II Depression
Keywords: bipolar disorder; depression; major depression; bipolar I depression; bipolar II depression; bipolar I disorder; bipolar II disorder; minocycline; minocin
MeSH Terms: conditions — Bipolar Disorder; Depression; Depressive Disorder, Major; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline (100 mg bid) will be administered as an adjunctive agent to conventional Health Canada-approved, or first-line CANMAT bipolar guideline-recommended, agents for bipolar disorder.
  Other Names: Minocin

SUMMARY:
Long-term studies have emphasized that depressive symptoms and episodes account for majority of the illness burden experienced by individuals with bipolar disorder (BD). Previous studies have shown that blood levels of proteins called pro-inflammatory cytokines are abnormal in individuals with bipolar depression. The investigators hypothesize that preventing the production or release of pro-inflammatory cytokines will result in improvement of depressive symptoms in individuals with bipolar depression. Minocycline is a medication that inhibits the activation of immune cells (i.e. microglia) in the brain and reduces the production of pro-inflammatory cytokines. Treatment with minocycline has been shown to have antidepressant-like effects in animal studies and improve symptoms of individuals with schizophrenia. In this study, minocycline (100 mg twice a day) will be administered for 8 weeks to determine if it is an efficacious antidepressant for individuals with bipolar depression.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is associated with a high-rate of non-recovery, recurrence, and inter-episodic dysfunction. Depressive symptoms and episodes dominate the longitudinal course of BD and differentially account for overall illness burden. During the past decade, substantial developments have been made in the pharmacological and psychosocial treatment of bipolar mania and maintenance, with relatively few treatments proven efficacious for bipolar depression. The absence of an explanatory disease model in bipolar disorder has limited the development and evaluation of genuinely novel agents for bipolar disorder.

Several lines of evidence implicate the inflammatory system as consequential and causative to mood disorder. Bipolar disorder is marked by alterations in inflammatory cytokines (e.g. TNF-alpha, IL-6). Moreover, pro-inflammatory activation in both healthy and medically ill individuals is associated with disturbances in affective, cognitive, and somatic function.

The clinical use of cytokine-based therapy has been demonstrated to induce and/or intensify affective symptomatology in non-psychiatric medical patients. Conventional pharmacological treatments (e.g. lithium) for bipolar disorder affects the production of pro-inflammatory cytokines as well as their gene expression. The encompassing aim of the study herein is to develop a novel treatment for bipolar depression based on a model of disease pathophysiology. Minocycline is a semisynthetic second-generation tetracycline, which exerts anti-inflammatory effects that are distinct from its antimicrobial properties.

Minocycline is a potent inhibitor of microglial activation and decreases expression of pro-inflammatory cytokines, chemokines and their receptors and suppresses the activity of matrix metalloproteinases. Minocycline has been shown to exert antidepressant-like properties in preclinical studies. Rats treated with minocycline monotherapy as well as combination treatment with an antidepressant (desipramine) exhibited significantly improved performance on the forced swim test. Adjunctive minocycline has been shown to be efficacious for the treatment of schizophrenia in a double-blind, randomized, placebo-controlled study. Subjects receiving minocycline exhibited a significant improvement in negative symptoms as well as global improvement as measured with the Clinical Global Impression (CGI). Significant improvement was also noted on measures of executive function, including executive function composite score, spatial recognition memory, cognitive planning, and intradimensional/extradimensional set shifting.

A total of 40 individuals between the ages of 18 and 65 meeting DSM-IV-TR criteria for a current major depressive episode as part of bipolar I or II disorder will be enrolled into an 8-week, open-label study with adjunctive minocycline (100 mg every 12 hours).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I or II disorder
* Meets criteria for a current major depressive episode
* A score of >= 20 on the HAMD-17 at the time of enrollment and at baseline
* Episode duration will be greater than 4 weeks but not longer than 12 months.

Exclusion Criteria:

* Insufficiently responding to >2 treatment strategies FDA/Health Canada-approved/guideline recommended for bipolar depression
* Acute manic or mixed episode
* An Axis I psychiatric disorder requiring primary clinical attention
* Clinically significant medical illness
* Treatment with minocycline or β-lactam antibiotics in the preceding 6 months
* Hypersensitivity to minocycline or any other tetracycline
* Physical injury requiring medical treatment or surgery in the last 6 months
* Pregnant or breast-feeding
* Inability to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 8 on the Montgomery Asberg Depression Rating Scale (MADRS) | Baseline, Week 1, 2, 4, 6, 8
  The MADRS assesses depressive symptoms

SECONDARY OUTCOMES:
Change from baseline to week 8 on the Hamilton Depression Rating Scale 17-item (HAMD-17) | Baseline, Week 1, 2, 4, 6, 8
  The HAMD-17 assesses depressive symptoms
Change from baseline to week 8 on the Somatic Symptom Inventory (SSI) | Baseline, Week 8
Change from baseline to week 8 on the Clinical Global Impression (CGI) Rating Scale | Baseline, Week 1, 2, 4, 6, 8
Change from baseline to week 8 in the in neurocognitive function | Baseline, Week 8
  California Verbal Learning Test- second edition (CVLT-II), Process Dissociation Task, Trail Making Test A and B, Verbal Fluency- Delis-Kaplan Executive Function System (D-KEFS,) Digit Symbol Substitution, Cognitive Failures Questionnaire
Monitoring of Side-effects from baseline to week 8 with the Toronto Side Effect Scale (TSES) | Week 1, 2, 4, 6, 8
Monitoring of suicide severity from baseline to week 8 with the Columbia Suicide Severity Rating Scale (C-SSRS). | Baseline, Week 1, 2, 4, 6, 8
Change from baseline to week 8 in concentrations of pro-and anti-inflammatory cytokines (e.g. TNFα, IL-1β, IL-2, IL-6, IL8, IFNγ, IL-4, IL-5, IL-10) | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Roger S McIntyre, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Levkovitz Y, Mendlovich S, Riwkes S, Braw Y, Levkovitch-Verbin H, Gal G, Fennig S, Treves I, Kron S. A double-blind, randomized study of minocycline for the treatment of negative and cognitive symptoms in early-phase schizophrenia. J Clin Psychiatry. 2010 Feb;71(2):138-49. doi: 10.4088/JCP.08m04666yel. Epub 2009 Nov 3. PMID 19895780
- [Background] Molina-Hernandez M, Tellez-Alcantara NP, Perez-Garcia J, Olivera-Lopez JI, Jaramillo-Jaimes MT. Antidepressant-like actions of minocycline combined with several glutamate antagonists. Prog Neuropsychopharmacol Biol Psychiatry. 2008 Feb 15;32(2):380-6. doi: 10.1016/j.pnpbp.2007.09.004. Epub 2007 Sep 14. PMID 17933448